CLINICAL TRIAL: NCT00886834
Title: A Randomized Control Trial of Misoprostol vs. Placebo Prior to IUD Insertion in Nulliparous Women
Brief Title: Misoprostol Prior to Intrauterine Device (IUD) Insertion in Nulliparous Women
Acronym: MPIIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24403
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2014-12-22 (Estimated); Status verified 2014-12

CONDITIONS: Contraception
Keywords: IUD insertion; Nulliparous women; Contraception; Family Planning; IUD insertion in nulliparous women
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Misoprostol (Experimental): Misoprostol 400 micrograms inserted vaginally or buccally, per the participants desire.
  Interventions: Drug: Misoprostol
- Placebo (Placebo Comparator): Pills which are identical to the study drug in appearance, taste, and smell.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Misoprostol — 400 micrograms inserted vaginally or buccally, per the participants desire prior to the IUD insertion.
  Other Names: Cytotec
  Arms: Misoprostol
Drug: Placebo — Pills which are identical to the study drug in appearance, taste, and smell.
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if inserting misoprostol in the vagina or between your cheek and gum before inserting an Intrauterine Device (IUD) in a woman who has never had a baby makes it easier and less painful.

DETAILED DESCRIPTION:
Intrauterine Devices (IUDs) are an excellent method of contraception but are underutilized in the U.S. IUD use is expanding in the U.S. and is now routinely recommended for nulliparous women. The cervix of a nulliparous woman has a smaller diameter and can lead to more difficult and uncomfortable IUD insertions. Because of misoprostol's known ability to cause cervical dilation, some family planning providers use this drug to facilitate insertion. While there is a wealth of data on the use of misoprostol prior to many procedures requiring cervical dilation there is minimal objective evidence assessing its effect on provider ease of insertion or patient comfort during IUD insertion in nulliparas. The goal of this project is to evaluate whether misoprostol relative to placebo prior to IUD insertion in nulliparous women eases insertion and decreases pain. The results of this trial will be contributed to a prospective meta-analysis on the subject.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* negative pregnancy test
* no prior pregnancies beyond 14 6/7 weeks
* no PID in last 3 months
* no current cervicitis
* be willing to follow-up in 1-2 months for an IUD string check.

Exclusion Criteria:

* active cervical infection
* current pregnancy
* prior pregnancy beyond 14 weeks gestation
* known uterine anomaly
* fibroid uterus distorting uterine cavity
* copper allergy/Wilson's disease (for Paragard)
* undiagnosed abnormal uterine bleeding
* cervical or uterine cancer.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD/MPH, Principal Investigator — University of Utah Department of Obstetrics and Gynecology
Locations (2):
- United States (2):
  - Planned Parenthood Association of Utah, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Swenson C, Turok DK, Ward K, Jacobson JC, Dermish A. Self-administered misoprostol or placebo before intrauterine device insertion in nulliparous women: a randomized controlled trial. Obstet Gynecol. 2012 Aug;120(2 Pt 1):341-7. doi: 10.1097/AOG.0b013e31825d9ec9. PMID 22825094
- [Derived] Turok DK, Espey E, Edelman AB, Lotke PS, Lathrop EH, Teal SB, Jacobson JC, Simonsen SE, Schulz KF. The methodology for developing a prospective meta-analysis in the family planning community. Trials. 2011 Apr 29;12:104. doi: 10.1186/1745-6215-12-104. PMID 21527040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from July 2009 to November 2010. All IUD insertions occurred at the University of Utah Ob/Gyn clinic.
Pre-assignment Details: Participants had an initial study visit where the consent was signed and they were given misoprostol or placebo to take at home. Participants and providers were blinded to the treatment group.
Period: Overall Study
Arm/Group | Misoprostol | Placebo
Started | 54 | 54
Completed | 54 | 51
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Misoprostol | Placebo | Total
Number analyzed (Participants) | 54 | 54 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 54 | 108
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.6 (3.8) | 24.8 (4.2) | 24.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 54 | 108
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 54 | 108

OUTCOME MEASURES:

1. Primary Outcome: Provider Perceived Ease of Insertion on a 100-point Visual Analogue Scale (VAS)
Description: VAS (anchors: 0 = extremely easy, 100 mm= impossible)
Time Frame: Immediately post IUD insertion
Population: 2 of the placebo patients received pre-medication for pain and were excluded and 1 of the placebo patients did not return for IUD insertion.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 54 | 51
units on a scale | 25.1 (3.5) | 27.4 (3.5)
Statistical Analysis 1: Comparison: Misoprostol vs Placebo; Test type: Superiority or Other; p = 0.64, t-test, 2 sided

2. Secondary Outcome: Patient Perceived Pain on a 100-point Visual Analogue Scale (VAS)
Description: VAS; anchors: 0 =none, 100 mm= worst imaginable
Time Frame: prior to insertion, immediately after insertion, and prior to clinic discharge
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Misoprostol | Placebo
Number analyzed (Participants) | 54 | 51
units on a scale
  prior to insertion | 17.1 (3.5) | 4.8 (2.0)
  immediately after insertion | 58.4 (3.3) | 56.9 (3.0)
  prior to clinic discharge | 35.1 (3.4) | 27.5 (2.4)

ADVERSE EVENTS:
Description: 2 of the placebo patients received pre-medication for pain and were excluded and 1 of the placebo patients did not return for IUD insertion.
Arm/Group | Misoprostol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/51
Other Adverse Events (participants affected / at risk) | 0/54 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No